CLINICAL TRIAL: NCT00471471
Title: Safety and Immunogenicity of Vaccination With Multi-Epitope Peptide Vaccine Containing MART-1, gp100, and Tyrosinase Peptides Given With the Combination of GMCSF and CpG Oligonucleotide (CpG 7909) in ISA-Oil Adjuvant for Patients With Recurrent Inoperable Stage III or Stage IV Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Recurrent Stage III or Stage IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahmad Tarhini (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ahmad Tarhini, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-173; NCI-2009-00159 (Registry Identifier: CTRP (Clinical Trials Reporting System)); PCI-IRB-0607048; CDR0000544402 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Intraocular Melanoma; Malignant Conjunctival Neoplasm; Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; iris melanoma; recurrent intraocular melanoma; metastatic intraocular melanoma; conjunctival melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Protein Subunit Vaccines; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peptide Vaccine + GM-CSF + Pfizer 3512676 in-ISA Oil (Experimental): The water-in-oil emulsion will consist of peptide (100 mcg/0.1 mL), GM-CSF (80 mcg/0.16 mL using lyophilized 500 mcg/vial reconstituted with 1 mL of sterile water), Pfizer PF3512676 (0.6 mg/0.04 mL using 15mg/mL vial) and 0.20 mLl of sterile saline.
  Vaccination will be given subcutaneously rotating truncal sites in the vicinity of the four nodal drainage groups of the four extremities, on days 1 and 15 of each cycle (1 cycle = 28 days) for a maximum of 13 cycles (1 year).
  Interventions: Biological: Peptide vaccine; Biological: GM-CSF; Biological: PF3512676

INTERVENTIONS:
Biological: Peptide vaccine — Multi-epitope peptide vaccine containing MART-1 (26-35, 27L), gp100 (209-217, 210M) and tyrosinase (368-376, 370D) peptides
Biological: GM-CSF — 80 mcg/0.16 mL using lyophilized 500 mcg/vial reconstituted with 1 mL of sterile water given subcutaneously rotating truncal sites in the vicinity of the four nodal drainage groups of the four extremities, on days 1 and 15 of each cycle (1 cycle = 28 days) for a maximum of 13 cycles (1 year).
  Other Names: Sargramostim
Biological: PF3512676 — 0.6 mg/0.04 mL given subcutaneously rotating truncal sites in the vicinity of the four nodal drainage groups of the four extremities, on days 1 and 15 of each cycle (1 cycle = 28 days) for a maximum of 13 cycles (1 year).
  Other Names: CpG 7909; agatolimod

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving vaccine therapy together with GM-CSF, CpG 7909, and incomplete Freund's adjuvant may make a stronger immune response and kill more tumor cells.

PURPOSE: This clinical trial is studying the side effects and how well vaccine therapy works in treating patients with recurrent stage III or stage IV melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of a peptide vaccine comprising MART-1:27-35 peptide, gp100:209-217 (210M) peptide, and tyrosinase peptide with sargramostim (GM-CSF) and CpG 7909 emulsified in incomplete Freund's adjuvant in patients with unresectable recurrent stage III or IV melanoma.
* Determine the efficacy of immunoadjuvants CpG 7909 and GM-CSF, in terms of a strong antigen-specific CD8+ T-cell response, in these patients.
* Determine the anti-pigmentary response to this regimen in these patients.
* Determine the anti-tumor response, in terms of objective tumor regression, progression-free survival, and overall survival, in patients treated with this regimen.

OUTLINE: This is a pilot study.

Patients receive peptide vaccine comprising MART-1:27-35 peptide, gp100:209-217 (210M) peptide, and tyrosinase peptide with sargramostim (GM-CSF) and CpG 7909 emulsified in incomplete Freund's adjuvant subcutaneously on days 1 and 15. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline, day 50-53, and day 91-94. Samples are examined by ELISPOT assay to measure lymphocyte immune response and by flow cytometry for biomarker quantification and T-cell response.

After completion of study treatment, patients are followed up periodically for at least 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma meeting the following criteria:

  * Unresectable recurrent disease
  * Stage III or IV disease
  * Cutaneous, ocular, or mucosal melanoma
* Measurable disease as defined by the RECIST criteria
* HLA-A2 positive
* Prior brain metastases allowed provided adequate surgical or radiologic treatment for brain disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* WBC ≥ 3,000/mm³
* Lymphocytes ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* Lactic dehydrogenase ≤ 2.0 times ULN
* aPTT < 40 seconds
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for ≥ 1 week before, during, and for ≥ 2 weeks after completion of study therapy
* No conditions of immunosuppression
* Negative titers for antinuclear antibody (≤ 1/80) and antidouble stranded DNA (≤ 1/10)
* No serious illnesses including, but not limited to, any of the following:

  * Bleeding disorders
  * Autoimmune diseases
  * Severe obstructive or restrictive pulmonary diseases
  * Active systemic infections
  * Inflammatory bowel disorders
* No serious cardiovascular disease including, but not limited to, any of the following:

  * Uncontrolled congestive heart failure
  * Hypertension
  * Cardiac ischemia
  * Myocardial infarction,
  * Severe cardiac arrhythmia
* HIV1 and 2 negative
* HTLV-1 negative
* Hepatitis B and C negative
* No significant psychiatric disease, medical intervention, or other condition that, in the opinion of the principal investigator, would limit study compliance
* No active infection within the past week, including unexplained fever (temperature > 38.1°C)

PRIOR CONCURRENT THERAPY:

* Fully recovered from prior major surgery
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas), hormonal therapy, radiotherapy, or biological therapy
* More than 1 week since prior antibiotics
* More than 28 days since prior investigational agent
* No prior vaccination with MART-1 (26-35, 27L), gp100 (209-217, 210M), and tyrosinase (368-376, 370D) peptides alone or in combination

  * Patients with history of vaccination with peptides other than MART-1 (26-35, 27L), gp100 (209-217, 210M), and tyrosinase (368-376, 370D) peptides allowed
* More than 4 weeks since prior and no concurrent systemic immunosuppressive therapy, including steroids

  * Patients on maintenance steroids given at physiologic doses because of adrenal insufficiency are eligible
* More than 2 weeks since prior and no concurrent treatment with systemic steroids, including oral steroids, continuous use of topical steroid creams or ointments, or any inhaled steroids
* No concurrent anticoagulants, except to keep an indwelling line patent
* No other concurrent anticancer therapy, including chemotherapy, immunotherapy, radiotherapy, experimental programs, and/or surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety | up to 1 year
  Number of grade 2 or greater allergic reactions (including generalized urticaria) or any grade 3 or greater adverse event

SECONDARY OUTCOMES:
Immunologic response | up to 94 days
  Change in the circulating effector T-cells.
Objective tumor regression | 2 months
  Change in tumor size will be performed at the end of cycle 2.
Depigmentation evaluation | up to 2 years
  Change in cutaneous depigmentation using careful inspection of the skin of the torso by a Wood's lamp.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad A. Tarhini, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Tarhini AA, Leng S, Moschos SJ, Yin Y, Sander C, Lin Y, Gooding WE, Kirkwood JM. Safety and immunogenicity of vaccination with MART-1 (26-35, 27L), gp100 (209-217, 210M), and tyrosinase (368-376, 370D) in adjuvant with PF-3512676 and GM-CSF in metastatic melanoma. J Immunother. 2012 May;35(4):359-66. doi: 10.1097/CJI.0b013e31825481fe. PMID 22495394